CLINICAL TRIAL: NCT00532545
Title: Bone Marker Changes In One Month Treatment With TERIPARATIDE (LY333334) Injections (rDNA Origin) in Men and Postmenopausal Women With Severe Osteoporosis
Brief Title: Bone Marker Changes With Teriparatide/Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6715; B3D-SU-S001
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Osteoporosis, Post-Menopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Teriparatide
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Teriparatide 20 micrograms/daily subcutaneously
  Other Names: LY333334

SUMMARY:
To test the hypothesis that Teriparatide injections given 20 micrograms/daily subcutaneously, for one month, are able to produce reliable changes in the bone marker in a severe osteoporotic population

ELIGIBILITY:
Inclusion Criteria:

* Presents with severe osteoporosis based on the disease diagnostic criteria and upon physician assessment
* Postmenopausal, nonpregnant, women older than 50 years of age, with previous fracture history such as hip, spine, wrist, ribs, clavicle, humerus, tibia, and fibula or men over 50 years of age with low impact fractures (fragility).
* Outpatients without concomitant diseases and with life expectancy of at least 3 years, according to the medical criteria.
* Cannot be on medicines that can disturb bone metabolism.
* Patients should be capable of self-injection, to learn the use of Pen device and are in agreement with its use.

Exclusion Criteria:

* Directly affiliated with the conduct of this study, or are the immediate family of someone directly affiliated with the conduct of this study (that is, Lilly employees, investigators, site personnel, or their immediate families). Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Received treatment within the last 30 days with a drug (not including study drug) that has not received regulatory approval for any indication at the time of study entry.
* Previously completed or withdrawn from this study or any other study investigating Teriparatide.
* Secondary osteoporosis or any disease that affects the bone metabolism, as renal osteodystrophy, osteomalacia, hypoparathyroidism, and hyperparathyroidism, and intestinal malabsorption.
* Cancer history in the 5 years prior to visit 1, with exemption of basocellular carcinoma treated and cervix carcinoma definitively treated at least 1 year before to visit 1

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-04; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that Teriparatide injections given 20 micrograms/daily subcutaneously, for one month, is able to produce reliable changes in the bone marker in a severe osteoporotic population in Puerto Rico.

SECONDARY OUTCOMES:
To test the hypothesis that this group of patients will have a high score in the survey used by IOF as an instrument to check risk factors.
Test the hypothesis that patients will have a high score in the survey used by IOF as an instrument to check risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Puerto Rico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fajardo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Humacao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com